CLINICAL TRIAL: NCT03468140
Title: A Matched Intervention Pilot Trial of Eculizumab Therapy to Reduce Preservation Injury in Human Macrosteatotic Liver Transplantation
Brief Title: Pilot Trial of Eculizumab Therapy to Reduce Preservation Injury in Human Macrosteatotic Liver Transplantation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to recruit due to COVID 19
Sponsor: Yale University (Other)
Collaborators: Ochsner Health System (Other); Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Sanjay Kulkarni, Associate Professor of Surgery (Transplant) and of Medicine (Nephrology), Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000021373
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: Five end-stage liver disease (ESLD) patients will be matched to 5 historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Current end stage liver disease patients (Experimental): Eculizumab
  Interventions: Drug: Eculizumab
- Historical controls (Other): The Ochsner database will be used to obtain 5 historical matches for each study participant. Matching criteria for each patient will include: 1) gender; 2) (MELD) Score ± 5; 3) age ± 5 years; 4) body mass index (BMI) ± 5 kg/m2; 5) donor macrosteatosis ± 5%; and 6) CIT± 3 hours.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Eculizumab — Eculizumab will be given at a dose of 1200mg diluted in 0.9% sodium chloride (NaCl) to 5mg/mL for a total volume of 240 mL administered by IV infusion over 25-45 minutes in the anhepatic-phase during the transplant procedure, and a second dose of 900mg diluted in 0.9% NaCl to 5mg/mL for a total volume of 180 mL administered by IV infusion over 25-45 minutes will be given 24 hours following the first dose.
  Arms: Current end stage liver disease patients
Other: No intervention — Historical control arm
  Arms: Historical controls

SUMMARY:
The number of liver transplants that can be performed is limited by the availability of organs. Livers that are steatotic (i.e., infiltrated by triglycerides and other fatty substances) are usually not used for transplants, due to increased risk of adverse events and deaths post-transplant. The investigators propose administering eculizumab to patients receiving macrosteatotic liver transplants and hypothesize that doing so will mitigate post-surgical adverse outcomes.

DETAILED DESCRIPTION:
Mortality from liver disease accounts for approximately 34,000-36,000 annualized deaths and represents 11.5 deaths per 100,000 persons in the United States(1). Liver transplant is the only established treatment for end-stage liver disease (ESLD) and advancements over the past decade have resulted in excellent long-term survival rates(2). Liver transplant is limited solely by organ availability, as the numbers of available organs for transplant has remained stagnant. Compounding this problem is the rising global public health problem of fatty liver disease, with projected increases in incidence of non-alcoholic liver disease (NASH), both in the West and in Asia(3). One potential source of liver grafts is donors with moderate to severe macrosteatosis, as grafts from these donors are routinely discarded due to greater associated patient morbidity and mortality(4-6). When these grafts are used for transplantation, the clinical metrics of preservation injury are directly correlated with the degree of steatosis(7). Steatotic liver grafts represent the single largest source of potential donor livers that currently remains unutilized and methods aimed at their successful use would directly lead to reduced mortality in patients with ESLD. Evidence from pre-clinical models indicates that complement-mediated mechanisms play a critical role in the pathogenesis of preservation injury, particularly in the presence of macrosteatosis(8, 9). Expansion of the donor pool using established, FDA-approved therapeutics that inhibit terminal complement offer an expedited and practical solution to this problem.

The investigators therefore hypothesize that complement activation downstream of C5 crucially mediates post-transplant liver allograft injury associated with preservation, ischemia and reperfusion (heretofore referred to as preservation injury) and that macrosteatosis enhances the graft's susceptibility to this complement-dependent injury. As a corollary, the investigators hypothesize that the anti-C5 mAb eculizumab will limit post-transplant preservation injury despite macrosteatosis, thereby decreasing early post-transplant liver dysfunction, and ultimately resulting in greater utilization of macrosteatotic livers for transplantation, with consequent reduction in mortality for patients with end-stage liver disease.

This study will test safety and efficacy of complement inhibition with eculizumab in the ESLD population receiving macrosteatotic liver transplants. The study will also determine if known associations of hepatic lipid metabolism and innate immune responses are mitigated under conditions of complement inhibition.

If an adverse reaction occurs during the administration of (IP), the infusion may be slowed or stopped at the discretion of the Investigator. If the infusion is slowed, the total infusion time should not exceed two hours. The adverse reaction will be considered an AE/SAE and needs to be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age>18, weight>40kg
* Recipients of first liver transplant
* Biopsy proven macrosteatosis of > or = 20%
* Cold ischemia time < 8 hours
* Recipients of brain-dead deceased donors

Exclusion Criteria:

* Dual organ transplants
* ABO incompatible
* Meningococcal vaccination refusal
* Dual barrier contraception refusal
* Recipients with acute liver failure
* Recipients with Hepatitis B or C viral loads
* Physiological MELD Score>35
* Donor liver biopsy showing combined Microsteatosis+Macrosteatosis>70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of Hepatocellular Injury | Days 1-7 following liver transplant.
  Hepatocellular injury will be assessed by aminotranferase (AST) that will be measured for 7 days following transplant.

SECONDARY OUTCOMES:
Alanine transaminase (ALT) recovery time | Days 1-7 following liver transplant.
  ALT will be measured for 7 days following transplant
Seven-day peak post-transplant (GCT) | Days 1-7 following liver transplant.
  GCT will be measured for 7 days following transplant
Gamma-glutamyl transpeptidase (GCT) recovery time | Days 1-7 following liver transplant.
  GCT will be measured for 7 days following transplant
International Normalized Ratio (INR) recovery time | Days 1-7 following liver transplant.
  INR will be measured for 7 days following transplant
Seven-day peak post-transplant creatinine | Days 1-7 following liver transplant.
  creatinine will be measured for 7 days following transplant

OTHER OUTCOMES:
One-year incidence of biopsy-proven acute transplant rejection | One year from date of transplant
Post-transplant blood loss | One year from date of transplant
One-year all-cause mortality | One year from date of transplant
One-year graft survival | One year from date of transplant
One-year all-cause infections | One year from date of transplant
One-year all-cause re-operation | One year from date of transplant
One-year all-cause hospital re-admission | One year from date of transplant
One-year biliary complications | One year from date of transplant
One-year vascular complications | One year from date of transplant

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kulkarni, M.D., Principal Investigator — Yale University
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States